CLINICAL TRIAL: NCT03749603
Title: A Study Assessing Iron Status and Anemia in Filipino School Children From MIMAROPA Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18.10.DAI
Record Dates: First submitted 2018-10-04; First posted 2018-11-21 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Intervention Model Description: Exploratory, interventional, one arm study
Masking Description: no masking required. assessments are both done on same subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIBAY meter (Experimental): Non-invasive measurement of red blood cell Zinc Protoporphyrin (ZnPP/haem ratio-µmol/mol haem) fluorescence in the microcirculation of the lower lip.
  Interventions: Device: TIBAY Meter

INTERVENTIONS:
Device: TIBAY Meter — fluorescence probe will be applied for 3-5 minutes onto the wet vermillion of the lower lip.

SUMMARY:
The purpose of this study is to assess the iron status and to confirm the usability of the non-invasive ZnPP measurement for screening the different stages of iron deficiency defined by standard measurements from blood.

DETAILED DESCRIPTION:
Brief description: The purpose of this study is to assess the iron status and to confirm the usability of the non-invasive ZnPP measurement for screening the different stages of iron deficiency defined by standard measurements from blood.

Detailed Description:

The primary objective of this study is to assess the iron status and the prevalence of the different stages of iron deficiency measured and defined by the standard blood iron measurements and by the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip.

The secondary objective is to compare and to assess the usability of the non-invasive ZnPP measurement versus other standard iron status measurements from blood in distinguishing the different stages of iron deficiency.

Subjects will be enrolled into the study after signing an assent form in addition to having parental informed consent signed. Total study duration is 1 day.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 - 11 years old
2. Having obtained his/her informed assent.
3. Informed consent signed by one parent or legal authorized representative if applicable.

Exclusion Criteria:

1. Subjects or subjects' parent(s) or legal representative who are not willing and not able to comply with scheduled visits and the requirements of the study protocol
2. Currently participating or having participated in another clinical trial within 4 weeks prior to trial start.
3. Any disease of the lip and mouth that does not allow performing the lip measurement.
4. Diagnosis of any blood disorders affecting red blood cells ( aplastic anemia, autoimmune hemolytic anemia, thalassemia)
5. Diagnosis of any blood disorders affecting white blood cells (lymphoma, multiple myeloma, myeloplastic syndrome)
6. Diagnosis of any blood disorders affecting platelets ( idiopathic thrombocytopenic purpura, primary thrombocythemia)
7. Diagnosis of blood plasma ( hemophilia, von Willebrand disease)
8. Diagnosis of acute or chronic inflammatory disease (respiratory tract, digestive tract -bowel, liver, and any kidney disease)
9. Diagnosis of any neoplastic disease

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1521 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Iron deficiency (ID stage I) | From Screening till study completion or up to 7 days, whichever comes first
  Iron status / prevalence of different stages of iron deficiency (ID) measured and defined by the standard blood iron measurements and the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip
Prevalence of Iron deficient erythropoiesis (ID stage II) | From Screening till study completion or up to 7 days, whichever comes first
  Iron status / prevalence of different stages of iron deficiency (ID) measured and defined by the standard blood iron measurements and the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip
Prevalence of iron deficiency anemia (ID stage III) | From Screening till study completion or up to 7 days, whichever comes first
  Iron status / prevalence of different stages of iron deficiency (ID) measured and defined by the standard blood iron measurements and the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip
Prevalence of Anemia but no ID | From Screening till study completion or up to 7 days, whichever comes first
  Iron status / prevalence of different stages of iron deficiency (ID) measured and defined by the standard blood iron measurements and the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip
Prevalence of Iron deficiency using total body iron stores (TBIS) | From Screening till study completion or up to 7 days, whichever comes first
  Iron status / prevalence of different stages of iron deficiency (ID) measured and defined by the standard blood iron measurements and the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip
Prevalence of iron deficiency using the non-invasive zinc protoporphyrin (ZnPP) measurements | From Screening till study completion or up to 7 days, whichever comes first
  Iron status / prevalence of different stages of iron deficiency (ID) measured and defined by the standard blood iron measurements and the non-invasive measurement of red blood cell Zinc Protoporphyrin fluorescence in the microcirculation of the lower lip

SECONDARY OUTCOMES:
Comparison the non-invasive ZnPP with other standard blood iron status measurements | From Screening till study completion or up to 7 days, whichever comes first
  Comparison the non-invasive ZnPP with other standard blood iron status measurements for (ferritin, soluble transferrin receptor, hemoglobin) By comparing accuracy/ sensitivity/ specificity/ positive predictive value/negative predictive value/ ROC curve

CONTACTS AND LOCATIONS:
Locations (1):
- Food and Nutrition Research Institute, City of Taguig, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Undecided